CLINICAL TRIAL: NCT00322647
Title: Cancer Center Trials: Reasons for Low Accrual Rates at One Academic Institution Vs. The Community Setting
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Claire Verschraegen, MD; Principal Investigator, University of New Mexico - CRTC
Other Study IDs: 4904C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2008-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. To identify reasons for low patient recruitment numbers to clinical trials in a cancer research center setting (and a community setting) in order to attempt to increase accrual rates.
2. To review the screening sheet for women who considered participating in the study of Tamoxifen and Raloxifene (STAR) for the prevention of breast cancer in high risk women through the University of New Mexico in Albuquerque from 1999 through 2004

DETAILED DESCRIPTION:
Objective 1: All new cancer patients seen for a four month period at the University of New Mexico Cancer Research and Treatment Center (UNM CRTC) (academic population) and for a six month-period at the New Mexico Cancer Care Alliance (NMCCA) (community setting). A careful screening log will be kept during this period with the research nurses cooperation in documenting 1) whether patients seen were accrued to a clinical trial, 2) what available trials the patient might possibly be eligible for, and 3) the reason for not registering on to a clinical trial.

Objective 2: To compare the responses to questions on the entry forms of those women who were eligible and declined participation to those who participated by Hispanic versus non-Hispanic ethnicity, we will access, copy, and analyze all the risk assessment profiles otherwise known as entry or eligibility forms completed by women who considered participating in the study of Tamoxifen and Raloxifene (STAR). Patterns of eligibility criteria and risk assessment will be described by ethnicity of women considered for entry into this chemopreventive randomized trial without the use of personal identifying data in accordance with the Health Insurance Portability Accountability Act of 1996 to maintain patient confidentiality

ELIGIBILITY:
Inclusion Criteria:

* Women who considered participating in the study of Tamoxifen and Raloxifene (STAR) for the prevention of breast cancer in high risk women through the University of New Mexico in Albuquerque from 1999 through 2004

Exclusion Criteria:

* Not specified.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-01; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States